CLINICAL TRIAL: NCT05108480
Title: Prospective and Multicenter Study to Assess the Safety and Effectiveness of a Physiotherapy Treatment Through Self-myofascial Release With Foam Roller in Patients With Hemophilic Knee Arthropathy: A Randomized Clinical Trial
Brief Title: Self-myofascial Release With Foam Roller in Patients With Hemophilic Knee Arthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: He-FoamKnee
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-myofascial release (Experimental): Each session will last approximately 15 minutes, with five physiotherapy sessions taking place over a period of 2 months. The Self-Myofascial release protocol for the lower limbs using a Foam Roller and and Solid Ball Massage, adapted to patients with hemophilic ankle arthropathy will include: Self-Myofascial release of the plantar region using and Solid Ball Massage; Release of the myofascial components of the back of the leg using a Foam Roller; Release of the myofascial components of the anterior part of the leg using a Foam Roller; Release of myofascial components of the hamstring region using a Foam Roller; Release of the myofascial components of the adductor muscles using a Solid Ball Massage in a sitting position; Release of the myofascial components of the abductor muscles using a Foam Roller in lateral decubitus; Release of the myofascial components of the pelvitrochanterian muscles using a Foam Roller in a sitting position.
  Interventions: Other: Experimental group
- Control group (No Intervention): The subjects included in the control group will not receive Physiotherapy sessions and will continue with their usual routine of activity and physical exercise, and with the same drug treatment schedule with FVIII / FIX and analgesic drugs.

INTERVENTIONS:
Other: Experimental group — This study followed the protocol designed for patients with hemophilic knee arthropathy. For its implementation, a 30-cm long15-cm diameter foam roller was used, and a ball 22 cm in length and 8 cm in diameter. The total duration of the intervention was 15 minutes, with 7 sessions per week over a period of 8 weeks. The physiotherapist who supervised the intervention followed up on all patients by telephone on a weekly basis to check for the absence of haemarthrosis during the intervention and to detect the possible need for protocol adaptations depending on the clinical situation of each patient. Each patient was individually provided with instructions as to how perform the exercises during the pretreatment evaluation, customizing the program if necessary. All patients had access to a mobile application, designed ad hoc for the research study (He-Foam®), where they could learn about the exercises through demonstration videos.
  Arms: Self-myofascial release

SUMMARY:
Introduction: Hemophilic ankle arthropathy is manifested by degenerative functional alterations (deficit of muscular strength, mobility and proprioception) (intra-articular alterations) and chronic pain. Myofascial release techniques are used to treat soft tissue adhesions, relieve pain, and reduce tissue sensitivity.

Design. A randomized clinical trial. Directed: To evaluate the safety and effectiveness of a myofascial self-release protocol with Foam Roller applied in patients with hemophilic knee arthropathy.

Patients: 58 patients with knee arthropathy will be recruited for inclusion in the study. The patients will be recruited in 5 centers, from different regions of Spain.

Intervention: Each session will last approximately 15 minutes, with five physical therapy sessions per week over a period of 8 weeks. Patients will be evaluated at the beginning of the study, after the intervention and after a follow-up period of 2 months. The treatment program includes 11 exercises to be administered bilaterally. A mobile application will be developed where each patient can observe the exercises to be performed.

Measurement instruments and study variables: digital goniometer (ankle range of motion); visual analog scale and pressure algometer (joint pain); Hemophilia Joint Health Score (Joint Condition); dynamometer evaluation (muscle strength); 6-minute walk test (lower extremity functionality); Mobile device (activity log); Finger floor test (muscle flexibility). At the same time, the study will make it possible to determine the joint bleeding caused by the applied physiotherapy treatment.

Expected results: demonstrate the safety of this physiotherapy technique in patients with hemophilia. Likewise, an improvement in ankle pain, function and joint movement is expected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a medical diagnosis of hemophilia A or B.
* Patients with a severe phenotype of hemophilia (<1% FVIII/FIX).
* Patients with a medical diagnosis of hemophilic knee arthropathy and more than 3 points on the Hemophilia Joint Health Score.
* Being over 18 years old.
* No scheduled orthopedic surgeries during the study phase

Exclusion Criteria:

* Patients with hemarthrosis in the month before the beginning of the study.
* Patients unable to walk.
* Severe functional alterations of the upper limb that prevented the exercises.
* Failure to sign the informed consent document

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline knee joint pain after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  Visual analogic scale (VAS). This scale will be used to evaluate the perception of joint pain, where knee joint pain ranges from 0 to 10 points (no pain to maximum perceived pain).

SECONDARY OUTCOMES:
Change from baseline knee pressure pain threshold after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  Pressure algometer. Measuring instrument used to evaluate pressure joint pain. The instrument shall consist of a measuring device attached to a hard rubber tip 1.1 cm in diameter. Its sphere shall be calibrated in kg/cm2 with divisions of 0.1 kg/cm2. The pressure algometry methodology applied was based mainly on the study by Hogeweg. Before taking the measurements, patients will be instructed to say "yes" as soon as pressure exerted by the algometer becomes slightly unpleasant. The pressure algometer shall be kept perpendicular to the surface of the skin with the right hand, stabilizing the axis of the instrument using the thumb and index finger of the left hand. The pressure shall be increased at a uniform rate of approximately 1 kg/cm2 per second. As soon as the subject, according to the instructions, says "yes", the pressure will be stopped and the score will be noted.
Change from baseline knee joint status after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  Hemophilia Joint Health Score (HJHS). This measuring instrument will be used to evaluate the joint condition of knees. It includes 8 items (inflammation and its duration, pain, atrophy and muscle strength, crepitus, and reduced flexion and extension) ranging from 0 to 20 points per joint (the higher the score, the greater the joint deterioration).
Change from baseline knee range of motion after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  Goniometry. Knee range of motion shall be measured using a goniometer. The assessment can be made with the patient standing. This measuring instrument allows more accurate measurements than those obtained with a universal goniometer
Change from baseline knee muscles strength after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  Dynamometry. The maximum isometric strength of the flexor and extensor muscles of the knee joint will be evaluated on both limbs with a manual dynamometer using a mark test. For this test, the rater needs to keep the dynamometer stationary while the patient exerts maximum force against it.
Change from baseline muscle flexibility after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  Fingertip-to-Floor Test. This test is used to assess the degree of flexibility of the posterior muscles of the lower limbs. This value is calculated as the distance between the fingertip and the floor when maximum hip flexion with knee extension is performed
Change from baseline of muscle activation of the quadriceps after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  Muscle activation of the quadriceps was evaluated with surface electromyography (surface electromyography model; Shimmer Sensing, Dublin, Ireland). Electrodes were placed accord-ing to the European recommendations for the use of surface electromyography. Bipo-lar rectangular silver/silver chloride (Ag/AgCl) electrodes were used, measuring 28 x 44 mm (Ambu® WhiteSensor 4200 model) with a 46 mm2 measurement area, 2 cm apart. For the patients to reach their maximum muscle strength, the rater provided the same verbal stimulus to motivate all the patients with each contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Murcia
Locations (1):
- University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No